CLINICAL TRIAL: NCT03304639
Title: A Randomized Phase II Study of Anti-PD1 Antibody [MK-3475 (Pembrolizumab)] Alone Versus Anti-PD1 Antibody Plus Stereotactic Body Radiation Therapy in Advanced Merkel Cell Carcinoma
Brief Title: Testing the Addition of Radiation Therapy to Immunotherapy for Merkel Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01817; NCI-2017-01817 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A091605 (Other: Alliance for Clinical Trials in Oncology); A091605 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2017-10-05; First posted 2017-10-09 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-09

CONDITIONS: Advanced Merkel Cell Carcinoma; Clinical Stage III Cutaneous Merkel Cell Carcinoma AJCC v8; Clinical Stage IV Cutaneous Merkel Cell Carcinoma AJCC v8; Metastatic Merkel Cell Carcinoma; Pathologic Stage III Cutaneous Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIA Cutaneous Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIB Cutaneous Merkel Cell Carcinoma AJCC v8; Pathologic Stage IV Cutaneous Merkel Cell Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (pembrolizumab) (Active Comparator): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab
- Group II (pembrolizumab, SBRT) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo SBRT for 3 doses during cycle 1.
  Interventions: Biological: Pembrolizumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Group II (pembrolizumab, SBRT)

SUMMARY:
This randomized phase II trial studies how well pembrolizumab with or without stereotactic body radiation therapy works in treating patients with Merkel cell cancer that has spread to other places in the body (advanced). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving pembrolizumab with stereotactic body radiation therapy may work better in treating patients with Merkel cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe the progression-free survival (PFS) of stereotactic body radiation therapy (SBRT) + pembrolizumab (MK-3475) compared to pembrolizumab (MK-3475) alone in advanced/metastatic Merkel cell carcinoma (MCC) patients.

SECONDARY OBJECTIVES:

I. To describe the PFS of SBRT + MK-3475 compared to pembrolizumab (MK-3475) alone across Response Evaluation Criteria in Solid Tumors (RECIST) measurable (including both radiated and non-radiated) cancer deposits.

II. To describe the overall response rate of SBRT + pembrolizumab (MK-3475) compared to pembrolizumab(MK-3475) alone in both radiated and in non-radiated deposit(s).

III. To determine the PFS at 6 months of SBRT + pembrolizumab (MK-3475) compared to pembrolizumab (MK-3475) alone across all cancerous deposits by RECIST.

IV. To determine the rate of grade > 3-4 adverse events, by organ system, by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

V. To determine the local control of SBRT treated tumors. VI. To calculate delivered radiation dose using cone-beam computed tomography (CT) images collected on the radiation treatment table in the final treatment position.

CORRELATIVE SCIENCE OBJECTIVES:

I. To test the utility of CT-based radiomics to predict radiation-induced pneumonitis and true delivered dose of SBRT based on cone beam collected imaging and diagnostic scans.

II. Biobanking for future correlative science projects.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo SBRT for 3 doses during cycle 1.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically (histologically or cytologically) proven diagnosis of MCC by local pathology review
* Have measurable disease based on RECIST 1.1 including at least two cancerous deposits; at least one deposit must be RECIST measurable while at least one deposit must meet criteria for SBRT; non-radiated tumor will be identified prior to randomization on the protocol
* Patients must have advanced or metastatic MCC defined as evidence of distant metastasis(es) on imaging

  * Patients with locoregionally confined disease are not eligible
* No prior immunotherapy for advanced/metastatic MCC
* Patients with known or suspected central nervous system (CNS) metastases, untreated CNS metastases, or with the CNS as the only site of disease are excluded; however, subjects with controlled brain metastases will be allowed to enroll; controlled brain metastases are defined as no radiographic progression for at least 4 weeks following radiation and/or surgical treatment (or 4 weeks of observation if no intervention is clinically indicated), and off of steroids for at least 2 weeks, and no new or progressive neurological signs and symptoms
* Patients having received palliative radiotherapy for extracranial metastasis(es) are eligible as long as there are 2 cancerous deposits that have not received prior radiation therapy (RT) and they meet the following criteria

  * No prior radiation therapy (> 5 Gy) to the metastasis intended to be treated with SBRT
* No history of the following:

  * Autoimmunity requiring systemic immunosuppression within 2 years
  * Patients known to be human immunodeficiency virus (HIV) positive are eligible if they meet the following:

    * CD4 counts >= 350 mm^3
    * Serum HIV viral load of < 25,000 IU/ml
* No other active malignancy that the investigator determines would interfere with the treatment and safety analysis
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown; therefore, for women of childbearing potential only, a negative (if your test schedule specifically indicates a urine or serum pregnancy test, add that information at this point) pregnancy test done =< 28 days prior to registration is required
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dl
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3.0 x upper limit of normal (ULN)
* Systolic blood pressure (BP) =< 150 mg HG
* Diastolic BP =< 90 mg HG
* Albumin > 3 mg/dl
* Blood urea nitrogen (BUN) =< 30 mg/dl
* Creatinine =< 1.7 mg/dl
* The following imaging workup to document metastases within 45 days prior to study registration are required: CT scans of the chest, abdomen and pelvis with radionuclide bone scan OR whole body (at least skull base to midthigh) positron emission tomography (PET)/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2026-09-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Luke, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (255):
- United States (255):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I (Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.>
  > Pembrolizumab: Given IV
- Group II (Pembrolizumab, SBRT): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo SBRT for 3 doses during cycle 1.> > Pembrolizumab: Given IV>
  > Stereotactic Body Radiation Therapy: Undergo SBRT
Period: Overall Study
Arm/Group | Group I (Pembrolizumab) | Group II (Pembrolizumab, SBRT)
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Pembrolizumab) | Group II (Pembrolizumab, SBRT) | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.0 (9.7) | 69.0 (9.2) | 72.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Will compare PFS in non-radiated lesion(s) of patients receiving either (a) stereotactic body radiation therapy (SBRT) + pembrolizumab compared to (b) pembrolizumab alone in patients with advanced Merkel cell carcinoma. Kaplan- Meier curves will be constructed and median PFS times will be calculated for each arm. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From randomization to either disease progression or death (without progression), assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Group I (Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  >
  > Pembrolizumab: Given IV
- Group II (Pembrolizumab, SBRT): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo SBRT for 3 doses during cycle 1.
  >
  > Pembrolizumab: Given IV
  >
  > Stereotactic Body Radiation Therapy: Undergo SBRT
Arm/Group | Group I (Pembrolizumab) | Group II (Pembrolizumab, SBRT)
Number analyzed (Participants) | 4 | 5
months | 7.5 [1.6 to NA] — Insufficient number of participants with events | 5.5 [3.7 to NA] — Insufficient number of participants with events

2. Secondary Outcome: PFS Among All Response Evaluation Criteria in Solid Tumors Lesions
Description: Same as the primary endpoint, but includes both irradiated and non-radiated lesions. It is a time to event endpoint and will be evaluated using the Kaplan- Meier method. Median PFS times will be calculated for each arm and a cox proportional hazards model will be constructed to determine if there is a PFS benefit for patients receiving SBRT + pembrolizumab compared to pembrolizumab alone.
Time Frame: From randomization to either evidence of disease progression or death (without evidence of progression), assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I (Pembrolizumab) | Group II (Pembrolizumab, SBRT)
Number analyzed (Participants) | 4 | 5
months | 7.5 [1.6 to NA] — Insufficient number of participants with events | NA [5.5 to NA] — Insufficient number of participants with events

3. Secondary Outcome: Overall Response Rate
Description: Defined as partial response (PR) on 2 consecutive evaluations. Response rates will be calculated and compared across treatment arms utilizing a chi-square test.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pembrolizumab) | Group II (Pembrolizumab, SBRT)
Number analyzed (Participants) | 4 | 5
Participants | 1 | 2

4. Secondary Outcome: Progression-free Survival
Description: The rates of success will be calculated and compared across treatment arms utilizing a chi-square test.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pembrolizumab) | Group II (Pembrolizumab, SBRT)
Number analyzed (Participants) | 4 | 5
Participants | 1 | 2

5. Secondary Outcome: Incidence of Adverse Events
Description: Graded according to National Cancer Institute's Common Terminology Criteria for Adverse Events, version 5.0. Maximum grade adverse events will be summarized by treatment arm in a tabular setting.
Time Frame: Up to 3 months
Reporting Status: Not Posted

6. Secondary Outcome: PFS for Lesions Chosen for Radiation Prior to Randomization
Description: The protocol irradiated tumors are considered to be controlled if they have no evidence of progression. No evidence of progression is defined as complete response, PR, or stable disease. Local control of the protocol-irradiated tumor will be described using the Kaplan-Meier technique.
Time Frame: Up to 3 years
Population: Group I did not receive radiation per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pembrolizumab) | Group II (Pembrolizumab, SBRT)
Number analyzed (Participants) | 0 | 5
Participants |  | 0

7. Secondary Outcome: Delivered Radiation Dose Using Cone-beam Computed Tomography (CT) Images
Description: Radiation doses will be summarized descriptively and compared to the planned dose.
Time Frame: Up to 3 years
Population: Group I did not receive radiation per protocol.
Measure: Median (Full Range); unit: cGY
Arm/Group | Group I (Pembrolizumab) | Group II (Pembrolizumab, SBRT)
Number analyzed (Participants) | 0 | 5
cGY
  Planned Dose Cycle 1 |  | 24 [8 to 24]
  Actual Dose Cycle 1 |  | 24 [8 to 24]
  Planned Dose Cycle 2: number analyzed (Participants) | 0 | 2
  Planned Dose Cycle 2 |  | 16 [8 to 24]
  Actual Dose Cycle 2: number analyzed (Participants) | 0 | 2
  Actual Dose Cycle 2 |  | 16 [8 to 24]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Group I (Pembrolizumab) | Group II (Pembrolizumab, SBRT)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Pembrolizumab) (N=4) | Group II (Pembrolizumab, SBRT) (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (28) | 1 (33)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (22) | 1 (8)
Blurred vision (Eye disorders) | 0 (0) | 1 (4)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (4)
Watering eyes (Eye disorders) | 0 (0) | 1 (8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (27)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (23)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (7)
Edema limbs (General disorders) | 1 (2) | 2 (28)
Fatigue (General disorders) | 1 (1) | 2 (59)
Fever (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (35)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (14)
Generalized edema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (5)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (4)
Wound infection (Infections and infestations) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (9) | 2 (2)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (3) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (21) | 1 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (6) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (35)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (35)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (11)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 2 (37)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (14)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (12)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (8)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (14)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (22)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3)
Hypertension (Vascular disorders) | 1 (1) | 1 (30)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Lymphedema (Vascular disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03304639/Prot_SAP_000.pdf